CLINICAL TRIAL: NCT03458286
Title: A Pilot Randomised Control Trial to Measure the Effectiveness of Combined Modulated Ultrasound and Electric Current Stimulation in Treating Diabetic Foot Ulcers
Brief Title: A Study Measuring the Effectiveness of Combined Modulated Ultrasound and Electric Current Stimulation as an Adjunctive Treatment in Treating Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Jagmed Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFUCUSECS
Record Dates: First submitted 2018-02-22; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcers; Chronic; Combined ultrasound and electric current stimulation; Adjunctive therapy
MeSH Terms: conditions — Diabetic Foot; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into an experimental arm and a control arm of the study. The experimental group will receive the adjunctive CUSECS treatment along their usual treatment for their diabetic ulcer twice weekly for 8 weeks using the BRH-A2 wound healing device. They will also have a follow up appointment 4 weeks after completion of treatment.
  The control group will be required to attend the diabetic foot clinic for their usual care for their diabetic foot ulcer with weekly review for a maximum of eight weeks. They will also have a follow up appointment 4 weeks after completion of treatment.
Who Masked: Outcomes Assessor
Masking Description: Analysis of data will be blinded and carried out by a statistician. Patient data will be coded and not identifiable directly. The key to the code book information will be secured separately from the dataset in an encrypted file, which will only be accessible by the researcher and the supervisors of the study. Therefore the each arm will be coded and none identifiable to the outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will be required to attend the diabetic foot clinic for their usual care for their diabetic foot ulcer with weekly review for a maximum of eight weeks. They will also have a follow up appointment 4 weeks after completion of treatment.
- Experimental Arm (Experimental): A device- BRH-A2 wound healing device will provide Combined ultrasound and electric current stimulation (CUSECS) treatment which is the intervention for this arm. Participants in this group will receive an adjunctive combined ultrasound and electric current stimulation (CUSECS) treatment along their usual treatment for their diabetic ulcer twice weekly for 8 weeks using the BRH-A2 wound healing device. They will also have a follow up appointment 4 weeks after completion of treatment.
  Interventions: Device: BRH-A2 wound healing device

INTERVENTIONS:
Device: BRH-A2 wound healing device — Combined ultrasound and electric current stimulation (CUSECS) is a combination therapy provided by the BRH-A2 wound healing device. This study is testing the effectiveness of the treatment CUSECS. The electric current stimulation is provided by attaching small electrodes around the ulcers. A probe is used on the ulcers to provide the ultrasound waves. Both aiming to increase the blood flow to an area to increase wound healing.
  Arms: Experimental Arm

SUMMARY:
The study aims to investigate if combined modulated ultrasound and electric current stimulation (CUSECS) is an effective adjunctive treatment to use to treat diabetic foot ulcers when compared against usual care. Consenting patients with diabetic foot ulcers (DFUS) and meet the inclusion criteria will be randomly allocated in to either an experimental group or a control group. The experimental group will receive the adjunctive CUSECS treatment along their usual treatment for their diabetic ulcer. They will be required to attend the Diabetic Foot clinic in St. James's hospital twice a week for a maximum of eight weeks. The CUSECS is provided by attaching small electrodes around the ulcers to provide electric current stimulation. A probe is used on the ulcers to provide the ultrasound waves. Both aiming to increase the blood flow to an area to increase wound healing. The control group will be required to attend the diabetic foot clinic for their usual care for their diabetic foot ulcer once a week for a maximum for eight weeks. Once a week both groups ulcers will be assessed and measured and a photograph solely of the wound will be taken for documentation of wound healing. Wound pain as determined using the 0-10 Numeric pain rating scale will also be measured once a week.

The movement in participant's ankle will be measured (flexion, extension, inversion) at the start and at the end of the study to see if treatment has improved its movement.

As part of this study participants' will also be requested to fill out a SF-36 questionnaire at the start and at the end of the 8 week trial. This questionnaire evaluates a person's health related quality of life in which the research wants to see if it is affected by a diabetic foot ulcer. The self-efficacy of participants will also be assessed using PROMIS® Item Bank v.1.0 - General Self-Efficacy at the start and at the end of the 8 week trial. The cost of treatment for each arm will be calculated taking into account both direct (cost of treatments, consumables etc.) and indirect costs (loss of earnings, travel, parking etc.). Therefore, as part of this study, participants will be asked about mode of transport and transport time to and from the clinic and if their diabetic foot ulcer has affected their ability to work.

Diabetic foot ulcer reoccurrence rates will be monitored in both groups by a follow up appointment 4 weeks after each group completes treatment or monitoring.

Data from both groups will be examined and compared to see if CUSECS is effective in healing DFUs. The primary outcome of interest is wound healing and is determined by the number of wounds healed and the time to complete wound healing within eight weeks. All data will be stored confidentially.

The study hypothesis is that there is be increased healing rates in subjects treated with CUSECS in combination with standard care compared to those treated with standard care alone.

This study aims to provide evidence for continuing improvement in treatment for those suffering with diabetic foot ulcers.

DETAILED DESCRIPTION:
Study Background:

Diabetes is predicted to be one of the greatest challenges for individuals and society as a whole into the future. Persons with diabetes are 50 times more likely to develop a foot ulcer than their non-diabetic counterparts (1). The prevalence of foot ulceration in this patient group is suggested to range from 3-10 %(1). These wounds are difficult to heal and this is often compounded by the presence of multiple co-morbidities. Furthermore, diabetes is the leading cause of non-traumatic limb amputation in the world (2). Within 18 months following amputation, almost 50 percent of these people will develop ulceration on the other limb and of these, 58% will have further amputations within three to five years(3). It is worthy of note that the three-year mortality rate after the first amputation is between 20 and 50 percent (4, 5). Having diabetes impacts negatively on the individuals' heath related quality of life when compared to the general population (6). The most important variable influencing changes in HRQOL is the presence of complications of diabetes. Having a foot ulcer causes a loss of mobility for the individual thereby decreasing social functioning. Furthermore almost 50% of people will suffer with intractable pain (6).

The International Working Group of the Diabetic Foot (IWGDF) highlight the continuing difficulties in selecting clinically effective treatments for diabetic foot infection and ulceration. In two commissioned systematic reviews they point to the large number of treatment options available while at the same time the relative weakness of evidence to support the use of many of these options (7, 8). Two of these treatments, electrostimulation and ultrasound, were utilised in this study. While both these technologies have been shown to be effective in chronic wound healing, the use of combined modulated ultrasound and electrical current stimulation (CUSECS) is a new and not widely studied treatment Avrahami (9). The merits of each treatment individually will be explored below.

Widespread interest and research into the use of electrostimulation is evident since the 1960s (10). Electrostimulation has been shown to have an effect on a range of mechanisms which are beneficial to wound healing including;

* Improvement of blood flow
* Improvement in tensile strength
* Stimulation of protein and DNA synthesis
* Reductions in oedema
* Decreased bacterial growth
* Promotion of epithelial, fibroblast, neutrophil and macrophage cells
* Reduction in pain. (11,12)

Peters, et al. carried out an RCT to assess the impact of a 50 V current being applied to the wounds of those in the intervention group overnight (8 hours) using a microcomputer. Both groups also received usual care. Results indicate that 65% healed in the treatment group treated vs 35% in the control group (p= 0.058). Wound size reduction was not statistically different between the groups and in both groups the more compliant patients had better outcomes (13).

Ultrasound has also shown promising results in the treatment of Diabetic foot ulcers (DFU). For example, Ennis, et al. with a sample of 133 patients treated the intervention group with 40 KHz of ultrasound at an intensity of 0.1 -0.5 W/cm2 as well as usual care. The treatment was administered 3 times a week for 4 minutes over 12 weeks or until healed. Results indicate a better healing rate in the intervention group than the control (40.7% vs 14.3% p = 0.0366) and the treatment was found to be well tolerated and had no ill effects (14). In a 3 armed study also with DFU patients Yao, et al. also applied treatments with low-frequency ultrasound. The three groups had differing amounts of ultrasound per week (Group 1: 3 x week, Group 2: 1 x week, Group 3: placebo). The 3 times per week group showed the greatest amount of wound size reduction compared with baseline (86% p < 0·05) leading the authors to conclude that the treatment applied when applied 3 times per week led to better wound outcomes (15).

The combination of these two treatments is not widely studied but given their potential and documented efficacy as outlined above the proposition to combine them would appear to be reasonable. Two published studies to date has looked at the combination of these therapies for DFUs (9). Avrahami et al. carried out a retrospective analysis of 300 wounds which were treated with CUSECS. They looked specifically at 65 wounds both diabetic foot ulcers (n=27) and venous leg ulcers (n= 38). Patients all had at least 8 treatments in a minimum of 4 weeks, twice weekly with CUSECS using the BRH-A2 device (BRH Medical). Results indicate that 59.3 % of the diabetic foot ulcers achieved 50% closure within 4 weeks. The authors found no significant association between gender, wound size on presentation or the longevity of the wound on the outcomes. In a small prospective case series O'Connor, et al. found a mean wound size reduction of 71% in DFUs when treated twice a week with CUSECS. They suggest that CUSECS offers promise as an adjunct therapy for diabetic foot ulcers (16). More comprehensive and robust evidence is now required to ascertain the effectiveness of CUSECS as a therapy for DFUs. This study aims to address that deficit.

This study's focus is to determine the impact of the use of CUSECS in DFUs. This study will build on the existing evidence and will provide the first RCT data for this therapy. It is envisaged that this can provide evidence for continuing improvement in treatment for those suffering with DFUs.

For this study the following protocol will be followed:

Number of Subjects Planned Sample sizes of 24-50 have been recommended for pilot feasibility studies (17-21). Therefore, a sample size of 46 will be selected for this study (23 per group), plus 10% to allow for dropout, giving a sample size of 50 evaluable participants (25 per group). An evaluable participant is one who satisfies all inclusion/exclusion criteria and who completes the study.

STANDARD OPERATING PROCEDURES

Recruitment and randomisation

Participants who attend the diabetic foot clinic in St. James's hospital who are interested in part taking in the study and who meet the inclusion criteria and who do not meet the exclusion criteria will be selected.

The podiatrist working in the diabetic foot clinic in each site will screen all subjects who express an interested in participating to ensure they meet the inclusion criteria and not the exclusion criteria.

The researcher will provide to the attending podiatrist a list of unique ID's with a corresponding randomised study group. The podiatrist will identify patients who meet the inclusion/exclusion study criteria and who are willing to participate in the study. If eligible, the podiatrist will issue the participant with either the control or experimental 'Patient Information Leaflet'. This allocation will be based on the systematic inclusion on the ID list. Subjects randomized to the experimental group will be identified by their randomization code beginning with A001 (for the first subject randomized to the experimental Group). Participants randomized to the control group will be identified by their randomization code beginning with B001 (for the first subject randomized to the control group) at this visit.

Informed Consent

Signed and dated written informed consent must be obtained from each patient prior to enrollment in the study.

The consent form must embody the requirements of informed consent as required by the Declaration of Helsinki and following the guidance provided in IE ISO 14155 (Appendix C). This consent form must have relevant Institutional Review Boards (IRB) / Ethical committee (EC) approval prior to use.

Signed (witnessed mark in the case of subjects who are unable to write) and dated informed consent must be obtained from each subject prior to enrollment in the study. Information on the trial will be offered both verbally and in written form to all potential subjects before informed consent is obtained. The investigator must explain to the patient the nature of the study, its purpose, procedures, expected duration, benefits and possible risks in participation.

This information will be offered in easy to understand non-technical language where possible. Subjects will be afforded ample time (not less than 24 hours) to consider whether or not to participate in the trial. The subject will be given the right to ask questions and be informed of their rights to withdraw from the study at any time without prejudice. A copy of the signed and dated informed consent form will be provided to the subject.

Study Schedule

Screening Visit

* The podiatrist working in the diabetic foot clinic in each site will screen all subjects who express an interested in participating to ensure they meet the inclusion criteria and not the exclusion criteria.
* The podiatrist will assign those subjects who meet the inclusion criteria with a unique ID provided by the investigator. This allocation will be based on the systematic inclusion on the ID list. They will issue them with relevant 'Patient information leaflet' to their randomisation group. This leaflet will contain background information on the study and the information on the relevant protocol and attendance requirements.
* These subjects will be screened by the study investigator to ensure that they do not meet any of the exclusion criteria.
* To ensure they meet the study eligibility criteria, medical history and demographics will be recorded and the ulcer will be assessed for any infection.
* The researcher will discuss the study information contained on the information leaflet with the potential participant, in a private room. This information will be provided in plain English and in a manner and pace that suits the individual.
* The researcher will inform the potential participant that they will meet with them at their next clinic visit to obtain consent (within a minimum of 24hours).

Assessment and treatment Visit

* The participant will attend their diabetic foot clinic in the hospital.
* The participant will be assisted by the study investigator and or the podiatrist in to a comfortable position on the patient plinth.
* Potential subjects will be rescreened for inclusion and exclusion criteria by the study researcher.
* All wound dressings will be removed by the study researcher or the clinic podiatrist. The foot ulcer will be assessed for signs of infection by the study researcher. Infection will be assessed clinically by signs and symptoms that include purulent drainage, erythema, warmth, cellulitis, increased exudation, malodor, increased tenderness or pain and fever.
* If a wound is considered infected by the researcher at the first visit, the subject will be excluded from participating in the trial. However, the subject can be rescreened for participation after complete resolution of the wound infection.
* Subjects who meet the inclusion criteria, have capacity to consent and wish to enroll on the study will be asked to sign and date the written informed consent form by the study researcher.
* If participants are unable to sign/ date or to make their mark on the consent form, this will be signed and dated by a witness.
* Subjects will be given a copy of the signed and dated consent form.
* Subjects randomized to the experimental group will be identified by their randomization code beginning with A001 (for the first subject randomized to the experimental group). They will continue their standard care with the addition of CUSECS twice a week for 8 weeks by the BRH-A2 device. A follow up appointment will be organised 4 weeks after receiving their last treatment.
* Subjects randomized to the control group will be identified by their randomization code beginning with B001 (for the first subject randomized to the control group) at this visit. These subjects will continue their standard care and will be monitored weekly for 8 weeks with a follow up appointment 4 weeks after their last review in clinic.
* Demographic and medical history information of subjects will be recorded in the Case Report Forms (CRFs) by the study researcher.
* At visit 1 the BRH-A2 documentation software will be opened on the BRH-A2 wound healing device by the study investigator and a specific participant file using the assigned randomization code will be set up on the system for each participant. Detailed patient data, including specific details regarding the location, type and characteristics of ulcer will be inputted. This file will be saved on the BRH-A2 system and will be used to store all participants relevant wound data for the duration of the trial. This data will be secured using the advanced privacy mechanisms which are inbuilt on the BRH-A2 wound healing device.
* Wound pain will be assessed, measured and recorded using the 0-10 Numeric pain rating scale.
* Quality of life score will be measured and recorded by the administration of the SF-36 questionnaire.
* Subjects will also be asked to fill out PROMIS® Item Bank v.1.0 - General Self-Efficacy questionnaire to assess their self-efficacy.
* Ankle Range of Motion of the foot with DFU will be measured in degrees using a goniometer for flexion, extension & inversion.
* Investigator assessment of the wound to include photograph and measurement using the BRH-A2 wound healing device integrated measurement technology will occur after any debridement if necessary has taken place and the wound is cleaned with normal saline (or other designated wound cleanser used within the clinic setting).
* Wound bed condition will be assessed using the Photographic Wound Assessment Tool (PWAT).
* For those in the experimental group, the first CUSECS treatment with the BRH-A2 wound healing device will be administered after all baseline evaluations have been completed. The following treatment process will be followed for the BRH-A2 treatment:

  * The participant will be given a clear explanation of the procedure and what to expect during the procedure.
  * The study investigator will apply the 4 electrode pads (disposable, single participant use) to clean dry skin around the target ulcer at a minimum distance of 5cm from the wound edges.
  * The BRH-A2 ultrasound probe will be covered with a clean single use liner. Ultrasonic waves are transmitted through a probe which is placed over the wound and the surrounding peri-wound.
  * The combined modulated ultrasound and electric current stimulation therapy will be applied for 15 minutes during each treatment. The present treatment parameters are set to deliver modulated frequency ultrasound of between 1.0-3.0MHz with a maximum intensity of 2.0W/cm². The BRH-A2 is present to deliver electric stimulation current frequencies of between 4000Hz - 4250Hz ±1 with inferential output waveforms and an interferential beat frequency of PPS 1-250Hz.
* Once all wound assessments and treatments are complete participants foot ulcers will be redressed according to their standard care treatment plan.
* Cost of treatment for each group will be recorded.
* The use of concomitant medications will be recorded on the Case Report Forms (CRFs).
* All adverse events will be recorded on the Case Report Forms (CRFs) and the SAE reporting forms if necessary at each visit.

Treatment period

Treatments will be scheduled for each group:

* Experimental group - twice weekly for 8 weeks (16 follow up visits and 1 final review at week 12)
* Control group- once weekly for 8 weeks (8 follow up visits and 1 final review at week 12)

The following will occur during treatment period:

* All wound dressings will be removed by the study researcher or clinic podiatrist. The foot ulcer will be assessed for signs of infection by the study investigator. Infection will be assessed clinically by signs and symptoms that include purulent drainage, erythema, warmth, cellulitis, increased exudation, malodor, increased tenderness or pain and fever.
* If a wound infection is detected during the trial, treatment with BRH-A2 will be discontinued and the subject will be treated according to the local hospital or clinic protocol for managing wound infection. Active treatment will resume once the infection has been resolved. If infection is present for more than 2 weeks, the subject will be discontinued from the study.
* The BRH-A2 documentation software will be opened on the BRH-A2 wound healing device and the relevant participant randomization coded file will be opened. Participant data will be updated on this file.
* Once a week for participants in both groups assessment of the wound through photograph and measurement using the BRH-A2 wound healing device integrated measurement technology will occur after any debridement if necessary has taken place and the wound is cleaned with normal saline (or other designated wound cleanser used within the clinic setting). Wound pain will be recorded using the 0-10 Numeric pain rating scale and Wound bed condition will be assessed using the assessed using the Photographic Wound Assessment Tool once a week also.
* CUSECS treatment with the BRH-A2 wound healing device will be administered to subjects in the experimental group as previously discussed twice a week.
* Once all wound assessments and treatments are complete the participant's foot ulcer will be redressed according to participant standard care treatment plan.
* Cost of treatment for each arm of the research will be recorded.

On the final visit for both groups:

* Wound pain will be assessed, measured and recorded using the 0-10 Numeric pain rating scale.
* Quality of life score will be measured and recorded by the administration of the SF-36 questionnaire.
* Subjects will also be asked to fill out PROMIS® Item Bank v.1.0 - General Self-Efficacy questionnaire to assess their self-efficacy.
* Ankle Range of Motion of the foot with DFU will be measured in degrees using a goniometer for flexion, extension & inversion.

  * The use of concomitant medications will be recorded on the Case Report Forms (CRFs).
  * All adverse events will be recorded on the Case Report Forms (CRFs) and the SAE reporting forms if necessary at each visit.
  * Throughout the process the treatment will be explained to the participants and they have the option to withdraw from the study at any time. They will be reassured that withdrawing from the study will not affect the treatment of their DFU by their podiatrist in the hospital.

Follow-up Assessments

Subjects who participated in the study will be followed up and reviewed 4 weeks after the final treatment. The following procedures will be conducted at the follow-up visit:

* Digital evaluation of wound surface area using BRH-A2 wound measurement software for any wounds that remain open or that have reopened.
* Assessment of participants' foot ulcers which remain open or have reopened. Photograph and measurement using the BRH-A2 wound healing device integrated measurement technology will occur once ulcers are exposed, debrided and are cleaned with normal saline (or other designated wound cleanser used within the clinic setting) as necessary.
* Wound bed condition will be assessed using the Photographic Wound Assessment Tool (PWAT).
* Wound pain will be assessed, measured and recorded using the 0-10 Numeric pain rating scale.
* Once all ulcer assessments and treatments are complete participants foot ulcers will be redressed with current standard care treatment plan if required.
* The use of concomitant medications will be recorded on the Case Report Forms (CRFs).
* All adverse events will be recorded on the Case Report Forms (CRFs) and the SAE reporting forms if necessary.
* Subjects will be discharged from the study. Duration of treatment

The total duration of the study for each subject will be 12 weeks:

* Experimental group: Twice weekly visits for 8 weeks (16 follow up visits and 1 final review at week 12).
* Control group: Once weekly visits for 8 weeks (8 follow up visits and 1 final review at week 12).

Withdrawals

Each participant will be informed that they have the right to withdraw study at any time and that this will not affect their treatment of their Diabetic foot ulcer (DFU). In addition, the investigator may discontinue a participant from the study at any time if the investigator considers it necessary for any reason including:

* Participant no longer meets inclusion/exclusion criteria.
* If the participant's physician for any reason instruct the withdrawal of the patient from the study.
* Adverse experiences, which include categories of intolerable side effects or current illnesses, that may preclude continued treatment or confound evaluation of the treatment outcome.
* If an infection is detected during the trial treatment with BRH-A2 will be discontinued. The subject must be temporarily withdrawn from the study. Active treatment can resume after the infection has been resolved. In this case the subject must start the study at Visit 1.
* If infection is present for more than 2 weeks, the subject will be discontinued from the study.
* Non-compliance with treatment regimen or study requirements
* Disease progression which requires results in inability to continue to comply with study procedures.
* Consent withdrawn.
* Patient fails to return for treatment up (after three documented attempts to contact the subject).
* An adverse event which results in inability to continue to comply with study procedures.

If a subject has not been withdrawn from the study and fails to return for their next scheduled visit during the 8 week trial, a good faith effort of 2 phone calls and 1 documented attempt will be made to contact the subject and determine the reason(s) why the subject failed to return for a necessary visit. The reason(s) for withdrawal must be recorded on the Case Report Form.

Data Analysis

Support from the Biostatistical Consulting and Support Services at the RCSI will be sought before undertaking statistical analyses.

Analysis Populations

Intent-to-Treat: All subjects who are randomized into the study following the pre-treatment period. However, any participant who withdraws with consent from the study have the right to withdraw their data up to the time of publication.

Per Protocol: All subjects who demonstrate compliance with the device treatment protocol by completing 80% of visits during the scheduled trial period (12 weeks).

Baseline Demographics and Patient Characteristics Subject demographics and baseline evaluations, including physical examination and medical history, will be summarized by analysis population using counts and percentages, as appropriate, for categorical variables (such as sex), and using means, standard deviations, medians, maxima, and minima, as appropriate, for continuous variables (such as age).

Statistical testing for baseline comparability between the treatment and control groups will be performed on variables that have the potential to influence CUSECS evaluations (such as ulcer size, ulcer duration, ulcer location, etc.).

Primary and Secondary Endpoints

The endpoint analyses will be conducted on the Per Protocol subject population. The primary endpoint will be the effectiveness of CUSECS on wound healing of DFUs as measured by the number of subjects with complete wound closure after 8 weeks of treatment and the time to reach complete wound closure. Difference in wound size - Percent difference in wound surface area will be recorded from baseline to subjects' final treatment (or sooner if complete wound healing occurs earlier.

The secondary endpoints are observational and not hypothesis driven. The efficacy analyses will be performed using descriptive statistics (e.g., arithmetic mean, standard deviation, frequency, etc.) for continuous and discrete variables, and graphical displays (e.g., tabulations, stem and leaf plots, etc.) of efficacy assessments will be generated, as appropriate.

Deviations from Statistical Plans

As appropriate, additional, exploratory analysis (e.g., regression by covariate) may be performed with data from this efficacy study. Any analysis of this type will be reported as exploratory.

Statistical Criteria for Study Termination

All reports of SAEs and UADEs will be evaluated by the study Principle Investigator (PI) and reported to the study site IRBs as required. The study may be suspended or terminated at any time without the need for statistical analysis by the investigator or the sponsor if the PI or any of the study IRBs determine that the BRH-A2 presents unacceptable risk to the study participants for reasons related to patient safety.

Ethics

The study will not be initiated until written approval has been obtained from the relevant Institutional Review Boards (IRB)/ Research Ethics Committee.

Throughout the study, data will only be identified by an identification number and the patient's initials. Jagmed Limited affirms and upholds the principle of the patient's right to protection against invasion of privacy. Throughout the study, data will only be identified by the randomization identification number.

Data Handling and Record Keeping

All data collected within this study is covered by Irish Law 'Data Protection Acts 1988 and 2003". All information collected during this study shall be kept strictly anonymously in keeping with the data protection acts.

A data management plan will be developed by the researcher before data collection commences. All data stored on the researcher's database will be protected with an encrypted password. Patient anonymity will be protected at all times as patient data will be coded and not identifiable directly. The key to the code book information will be secured separately from the dataset in an encrypted file, which will only be accessible by the researcher and the supervisors of the study.

A password protected folder will be set up on the RCSI V: DRIVE which will be used to store electronic data securely. All hard copy data will be scanned electronically and saved in the secure V: DRIVE folder. Hard copy data will be shredded once scanned and saved on the V:Drive folder. All research subject data stored on the BRH-A2 device will be backed up onto the secure V:Drive folder. Research data will be stored for a period of 5 years in compliance with the Data Protection Acts 1988 and 2003.

Quality Control and Quality Assurance

"The sponsor is responsible for implementing and maintaining quality assurance and quality control systems with written SOPs to ensure that trials are conducted and data are generated, documented (recorded) and reported in compliance with the protocol, GCP, and the applicable regulatory requirement (s)."

"Monitors should be appointed by the sponsor. The monitor should be appropriately trained and have the scientific and/or clinical knowledge needed to monitor the trial adequately."

"The purpose of trial monitoring is to verify that:

* The rights and well-being of human subjects are protected.
* The reported trial data are accurate, complete, and verifiable from source documents.

The conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with the applicable regulatory requirement(s) (22).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a diagnosed diabetic.
* Participants who have the capacity to provide informed consent prior to participation in the study.
* Participants must be aged 18 or over on the day of the informed consent.
* Participants have an ulcer that has been present for at least 60 and less than 365 days.
* Participants and/or caregiver must be willing and able to comply with all study procedures and scheduled follow-up visits, for the duration of the study.

Exclusion Criteria:

* Subjects without capacity to consent or those who do not provide informed consent.
* Ulcers that have a total surface area greater than 15 cm2 as measured by a member of the study staff.
* Unwilling to continue with their standard wound care therapy for the study duration.
* Clinical evidence of infection or gangrene on any part of the affected foot or leg. A subject with clinically infected wound(s) who otherwise meets the study criteria may enter the study after successful treatment of the for wound infection.
* Target ulcer involving exposure of tendon, bone or joint capsule, or any tunnelling or sinus tracts (it is acceptable to have ulcers extending through the dermis and into subcutaneous tissue with presence of granulation tissue).
* Target ulcer treatment with a wound dressing containing human growth factors, engineering tissues, or skin substitutes (e.g. Apligraf, Dermagraf, Regranex etc) within 30 days of screening visit or planned during the study duration.
* History of bone cancer or metastatic disease of the affected limb, radiation therapy to the affected limb, or chemotherapy within the 12 months prior to screening visit.
* Suspected or confirmed malignancy of the wound.
* Participation in another drug or device study for the treatment of diabetic foot ulcer within 30 days of screening visit.
* Vascular procedures performed within 30 days of screening visit.
* Active bleeding tissue or untreated haemorrhagic conditions.
* Active or suspected DVT or thrombophlebitis.
* Conditions which, in the judgment of the treating investigator, may severely compromise the subject's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Total wound healing | 8 weeks
  The number of wounds that completely heal in the experimental group compared to control group. This may be presented in either or both following formats:
  * The proportion of wounds completely healed (frequency of complete healing by group).
  * The time to complete wound healing.

SECONDARY OUTCOMES:
Changes in wound bed condition. | 8 weeks
  Wound bed condition will be assessed using the Photographic Wound Assessment Tool (PWAT)
Patient reported quality of life | 8 weeks
  The effect of a DFU on a person's health related quality of life will be evaluated through SF-36 questionnaire.
Wound pain | 8 weeks
  Wound pain as determined using the 0-10 Numeric pain rating scale (NPRS). The NPRS is an 11-point scale from 0-10 with "0" indicating no pain and "10", the most intense pain imaginable. Patients verbally select a value that is most in line with the intensity of pain that they are experiencing.
Self-efficacy | 8 weeks
  Identifying patient self-efficacy will be carried out using the PROMIS® Item Bank v.1.0 - General Self-Efficacy
Cost of treatment per arm (economic analysis direct cost and in-direct costs). | 8 weeks
  Cost of treatment for each arm of the research will be monitored and calculated taking into account both direct (cost of treatments, consumables etc.) and indirect costs (loss of earnings, travel, parking etc.).
Ankle Range of Motion | 8 weeks
  Ankle Range of Motion will be measured in degrees using a goniometer for flexion, extension & inversion
Diabetic foot ulcer reoccurrence rates | 4 weeks after the treatment trial is completed (16 weeks)
  Diabetic foot ulcer reoccurrence rates will be monitored in both groups by a follow up appointment 4 weeks after each group completes treatment or monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Tom O' Connor, DR., Principal Investigator — Royal College of Surgeons in Ireland; Declan Patton, DR, Principal Investigator — Royal College of Surgeons in Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteiro-Soares M, Boyko EJ, Ribeiro J, Ribeiro I, Dinis-Ribeiro M. Predictive factors for diabetic foot ulceration: a systematic review. Diabetes Metab Res Rev. 2012 Oct;28(7):574-600. doi: 10.1002/dmrr.2319. PMID 22730196
- [Background] Dubsky M, Jirkovska A, Bem R, Fejfarova V, Skibova J, Schaper NC, Lipsky BA. Risk factors for recurrence of diabetic foot ulcers: prospective follow-up analysis in the Eurodiale subgroup. Int Wound J. 2013 Oct;10(5):555-61. doi: 10.1111/j.1742-481X.2012.01022.x. Epub 2012 Jun 19. PMID 22712631
- [Background] Apelqvist J. Diagnostics and treatment of the diabetic foot. Endocrine. 2012 Jun;41(3):384-97. doi: 10.1007/s12020-012-9619-x. Epub 2012 Feb 25. PMID 22367583
- [Background] Apelqvist J, Larsson J. What is the most effective way to reduce incidence of amputation in the diabetic foot? Diabetes Metab Res Rev. 2000 Sep-Oct;16 Suppl 1:S75-83. doi: 10.1002/1520-7560(200009/10)16:1+3.0.co;2-8. PMID 11054894
- [Background] Kuehn BM. Prompt response, multidisciplinary care key to reducing diabetic foot amputation. JAMA. 2012 Jul 4;308(1):19-20. doi: 10.1001/jama.2012.6778. No abstract available. PMID 22760271
- [Background] Winkley K, Sallis H, Kariyawasam D, Leelarathna LH, Chalder T, Edmonds ME, Stahl D, Ismail K. Five-year follow-up of a cohort of people with their first diabetic foot ulcer: the persistent effect of depression on mortality. Diabetologia. 2012 Feb;55(2):303-10. doi: 10.1007/s00125-011-2359-2. Epub 2011 Nov 6. PMID 22057196
- [Background] Game FL, Apelqvist J, Attinger C, Hartemann A, Hinchliffe RJ, Londahl M, Price PE, Jeffcoate WJ; International Working Group on the Diabetic Foot. Effectiveness of interventions to enhance healing of chronic ulcers of the foot in diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:154-68. doi: 10.1002/dmrr.2707. PMID 26344936
- [Background] Peters EJ, Lipsky BA, Aragon-Sanchez J, Boyko EJ, Diggle M, Embil JM, Kono S, Lavery LA, Senneville E, Urbancic-Rovan V, Van Asten SA, Jeffcoate WJ; International Working Group on the Diabetic Foot. Interventions in the management of infection in the foot in diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:145-53. doi: 10.1002/dmrr.2706. PMID 26344844
- [Background] Avrahami R, Rosenblum J, Gazes M, Rosenblum S, Litman L. The Effect of Combined Ultrasound and Electric Field Stimulation on Wound Healing in Chronic Ulcerations. Wounds. 2015 Jul;27(7):199-208. PMID 26192738
- [Background] Junger M, Arnold A, Zuder D, Stahl HW, Heising S. Local therapy and treatment costs of chronic, venous leg ulcers with electrical stimulation (Dermapulse): a prospective, placebo controlled, double blind trial. Wound Repair Regen. 2008 Jul-Aug;16(4):480-7. doi: 10.1111/j.1524-475X.2008.00393.x. PMID 18638265
- [Background] Kloth LC. Electrical Stimulation Technologies for Wound Healing. Adv Wound Care (New Rochelle). 2014 Feb 1;3(2):81-90. doi: 10.1089/wound.2013.0459. PMID 24761348
- [Background] Kloth LC. Electrical stimulation for wound healing: a review of evidence from in vitro studies, animal experiments, and clinical trials. Int J Low Extrem Wounds. 2005 Mar;4(1):23-44. doi: 10.1177/1534734605275733. PMID 15860450
- [Background] Peters EJ, Lavery LA, Armstrong DG, Fleischli JG. Electric stimulation as an adjunct to heal diabetic foot ulcers: a randomized clinical trial. Arch Phys Med Rehabil. 2001 Jun;82(6):721-5. doi: 10.1053/apmr.2001.23780. PMID 11387573
- [Background] Ennis WJ, Foremann P, Mozen N, Massey J, Conner-Kerr T, Meneses P. Ultrasound therapy for recalcitrant diabetic foot ulcers: results of a randomized, double-blind, controlled, multicenter study. Ostomy Wound Manage. 2005 Aug;51(8):24-39. PMID 16234574
- [Background] Yao M, Hasturk H, Kantarci A, Gu G, Garcia-Lavin S, Fabbi M, Park N, Hayashi H, Attala K, French MA, Driver VR. A pilot study evaluating non-contact low-frequency ultrasound and underlying molecular mechanism on diabetic foot ulcers. Int Wound J. 2014 Dec;11(6):586-93. doi: 10.1111/iwj.12005. Epub 2012 Nov 19. PMID 23163982
- [Background] O'Connor, T. et al. in EWMA (Amsterdam, 2017).
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Julious, S. A. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics 4, 287-291, doi:10.1002/pst.185 (2005).
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] RCSI (2017) Introduction to Clinical Research and Good Clinical Practice Including Integrated Addendum to GCP Guidelines (E6 (R2) Version 4